CLINICAL TRIAL: NCT02328196
Title: Validation of a Revised Version of the Danish McGill Ingestive Skills Assessment for Measuring Dysphagic Clients' Performance During Meals
Brief Title: Validation of a Revised Version of the Danish McGill Ingestive Skills Assessment
Status: Completed | Type: Observational
Sponsor: Metropolitan University College (Other)
Responsible Party: Principal Investigator, Tina Hansen, Assistant professor, PhD, Metropolitan University College
Other Study IDs: MetropolitanUC
Record Dates: First submitted 2014-12-17; First posted 2014-12-31 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Deglutition Disorders
Keywords: Outcome and Process Assessment (Health Care); Rasch analysis; Meal time performance
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: The Danish McGill Ingestive Skills Assessment (MISA-DK) — The MISA measures the performance of dysphagic patients during the patient's usual mealtime routine.

SUMMARY:
The McGill Ingestive Skills Assessment (MISA) for measuring dysphagic clients' functional performance during meals has been previously translated into Danish (MISA-DK) and this translated version validated. Critical issues about the construct validity of the scale, per se, had been raised. Consequently, major revisions of the MISA-DK have been undertaken, which necessitates a new validation process. Therefore, the purpose of this study is to evaluate the construct validity of a revised version of the MISA-DK when used amongst dysphagic adults in hospitals settings and community services.

DETAILED DESCRIPTION:
This study will assess the construct validity of a revised version of MISA-DK in the acute and rehabilitative settings by testing it for fit against a multidimensional Rasch model.

Participants in this research will be 500 dysphagic clients from several centres in Denmark, namely 250 acute patients from three Danish Regional university Hospitals in Herning, Hjørring and Odense, and 250 clients in the rehabilitation setting from the Århus Rehabilitation Institute, Hillerød Rehabilitation Institute and the Rehabilitation division of Copenhagen.

Participants who are judged to have a swallowing problem are assessed with the MISA-DK by special educated occupational therapists The MISA-DK assessment are implemented as a part of the usual assessment routine at the occupational therapy departments at the included centres and will be administered immediately after referral to Occupational therapy. This research will be the first to implement and assess a standardised method for assessing mealtime performance for dysphagia in dysphagic patients across the continuum of diagnosis and rehabilitation recovery.

The application of the Multidimensional Rasch models to the MIS-DK data aims to identify the combination of items in the MISA-DK that provide the highest level of specific objectivity and statistical sufficiency when determining ingestive skill ability. Furthermore, Differential item function by diagnosis, age and setting will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of swallowing difficulties associated with aging and/or previous or current diagnosis of, but not limited to head and neck cancer (treatment may include surgery, radiation or chemotherapy, or a combination of more than one), stroke, cervical spine abnormality, brain tumor, cardiovascular surgery, Parkinson's disease or multi-morbidity.

  * Fulfils five criteria for direct swallowing evaluation: able to remain alert for at least 15 minutes; able to sit in a chair or bed in at least a 60° upright position, able to swallow saliva, able to cough voluntarily, able to clear the throat twice.
  * Have the capacity to provide informed consent.

Exclusion Criteria:

* The clients are excluded in case of: no dysphagia, known severe cognitive impairment, terminally illness (predicted survival less than 6 months), known contraindications to ingest foods or liquids, poorly controlled psychosis, inability to read consent form; inability or unwillingness to give written informed content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clients +18 years referred to occupational therapy for swallowing evaluation because of known or suspected dysphagia
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Danish version of The McGill Ingestive Skills Assessment (MISA-DK) | 1 year
  The MISA-DK is administered as observation of dysphagic clients performance during a usual meal with 14 different textures (four liquids and ten solids). The MISA-DK is composed of 36 ingestive skill items distributed into four subscales: positioning for meals (four items); self-feeding skills, judgment and behavior (seven items); and oral motor skills for liquid (11 items) and solid ingestion (14 items). All items are scored on a three-point ordinal scale (1=absent ingestive skill; 2=insufficient ingestive skill performance; 3=adequate ingestive skill performance), which are summated into a total score. The scores of the 36 ingestive skill items serve as a basis for rehabilitation planning and diet recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Hansen, PhD, Principal Investigator — Metropolitan University College
Locations (1):
- Tina Hansen, Copenhagen, N, Denmark

IPD SHARING:
Plan to Share IPD: No
Individuel participant data are not available for other than the principal Investigator. This is approved by the Danish Data Protection Authority.